CLINICAL TRIAL: NCT07241819
Title: Evaluate the Efficacy and Safety of Ivonescimab Monotherapy or in Combination With Chemotherapy as Neoadjuvant/Adjuvant Therapy for Resectable Non-small Cell Lung Cancer
Brief Title: Ivonescimab Monotherapy or in Combination With Chemotherapy as Neoadjuvant/Adjuvant Therapy for Resectable Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wu Nan, Professor, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ75-ZY01
Record Dates: First submitted 2025-07-20; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: II-IIIB (T3N2) Resectable Non-small Cell Lung Cancer; Perioperative
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm1 PD-L1 TPS≥50% (Experimental)
  Interventions: Combination Product: Ivonescimab/surgery
- Arm2 PD-L1 TPS≥50% (Active Comparator)
  Interventions: Combination Product: Ivonescimab/chemotherapy/surgery
- Arm3 PD-L1 TPS<50% (Experimental)
  Interventions: Combination Product: Ivonescimab/chemotherapy/surgery
- Arm4 PD-L1 TPS<50% (Active Comparator)
  Interventions: Combination Product: Ivonescimab/chemotherapy/surgery

INTERVENTIONS:
Combination Product: Ivonescimab/surgery — Ivonescimab monotherapy (4 cycles)→surgery→Ivonescimab(13 cycles)
  Arms: Arm1 PD-L1 TPS≥50%
Combination Product: Ivonescimab/chemotherapy/surgery — Ivonescimab + 1cycle of platinum-based chemotherapy followed by 3 cycles of Ivonescimab monotherapy→surgery→Ivonescimab(13 cycles)
  Arms: Arm3 PD-L1 TPS<50%
Combination Product: Ivonescimab/chemotherapy/surgery — Ivonescimab + platinum-based chemotherapy (4 cycles)→surgery→Ivonescimab(13 cycles)
  Arms: Arm2 PD-L1 TPS≥50%
Combination Product: Ivonescimab/chemotherapy/surgery — Ivonescimab + platinum-based chemotherapy (4 cycles)→surgery→Ivonescimab(13 cycles)
  Arms: Arm4 PD-L1 TPS<50%

SUMMARY:
This study is a prospective, II Phase clinical trial designed to evaluate the efficacy and safety of ivonescimab as monotherapy or in combination with platinum-based chemotherapy in the perioperative treatment of resectable non-small cell lung cancer (NSCLC).

Patients are stratified by PD-L1 expression level (TPS ≥50% vs. <50%) and randomized in a 2:1 ratio to differentiated neoadjuvant treatment arms: PD-L1≥50% subgroup: Ivonescimab monotherapy (4 cycles) vs. ivonescimab + platinum-based chemotherapy (4 cycles); PD-L1<50% subgroup: Ivonescimab + 1 cycle of chemotherapy followed by 3 cycles of monotherapy vs. ivonescimab + platinum-based chemotherapy (4 cycles). All patients subsequently receive 13 cycles of ivonescimab as adjuvant maintenance therapy postoperatively.

As the first study to explore a PD-L1-directed chemotherapy de-escalation strategy, this trial aims to reduce treatment toxicity while maintaining efficacy, thereby providing a novel personalized precision therapy pathway for resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form;
2. Aged ≥ 18 years and ≤ 75 years , both males and females are eligible;
3. ECOG PS score of 0 or 1;
4. Patients with non-small cell lung cancer confirmed by histopathology or cytology, and with resectable clinical stage II-IIIB (T3N2) (according to the 8th edition of lung cancer TNM staging by the Union for International Cancer Control and the American Joint Committee on Cancer);
5. No prior anti-tumor treatment has been received;
6. No known EGFR sensitive mutations/ALK gene translocations;

Exclusion Criteria:

1. Patients with large cell carcinoma, mixed-cell lung cancer, or those with small cell lung cancer components in the mixture;
2. Presence of locally advanced unresectable or metastatic disease;
3. Palliative local treatment for non-target lesions within 2 weeks before the first administration; receipt of non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 used for the treatment of thrombocytopenia) within 2 weeks before the first administration; receipt of Chinese herbal medicines or proprietary Chinese medicines with anti-tumor indications within 1 week before the first administration.
4. Severe infection occurred within 4 weeks before the first administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection treated with systemic anti-infective therapy within 2 weeks before the first administration (excluding antiviral therapy for hepatitis B or hepatitis C);
5. Major surgical operation or severe trauma occurred within 4 weeks before the first administration, or those with a plan for major surgical operation within 4 weeks after the first administration (determined by the researcher); minor local surgery performed within 3 days before the first administration (excluding peripherally inserted central catheterization and venous access port implantation);
6. History of severe bleeding tendency or coagulation dysfunction; presence of clinically significant bleeding symptoms within 1 month before the first administration, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or expectorating ≥ 1 teaspoon of fresh blood or small blood clots, or coughing up only blood without sputum; those with blood-tinged sputum are allowed to enroll), nasal bleeding (excluding epistaxis and retrograde epistaxis); receipt of continuous antiplatelet or anticoagulant therapy within 10 days before the first administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response（pCR）rate | At the time of postoperative pathological assessment，Up to approximately 2 years
  pCR is defined as the proportion of subjects who have completed surgery and, after the completion of neoadjuvant therapy, have no residual tumor in the resected primary tumor site and lymph nodes as evaluated by local pathology experts.

SECONDARY OUTCOMES:
Major Pathological response，MPR | At the time of postoperative pathological assessment，Up to approximately 2 years
  MPR is defined as the proportion of patients who have completed surgery and, as evaluated by local pathology experts, have residual viable tumor cells accounting for ≤10% in the resected primary tumor foci and lymph nodes.
R0 resection rate | At the time of postoperative pathological assessment，Up to approximately 2 years
  the proportion of patients who have completed surgery and achieved a pathological complete resection of the primary tumor, as evaluated by the researchers and local pathology experts.
Objective Response Rate，ORR | After completion of neoadjuvant therapy and before surgery，Up to approximately 2 years
  the proportion of patients whose tumor volume reduction meets the pre-specified criteria (complete response/partial response, CR/PR) and can be maintained for the minimum required duration in accordance with recognized response evaluation criteria (such as RECIST version 1.1 for solid tumors)
24 months Event-Free Survival（EFS）% | At 24 months after the first administration of study drug to the subjects
  the time from the first administration of the drug in the Full Analysis Set (FAS) to the occurrence of any of the following events, whichever comes first: disease progression evaluated according to RECIST v1.1, local recurrence, distant metastasis, or death from any cause.
incidence rate of adverse events | Up to approximately 2 years

OTHER OUTCOMES:
Explore biomarkers in subjects' tumor tissues that predict the efficacy of evosimab | Up to approximately 2 years
Explore biomarkers in subjects' blood that predict the efficacy of evosimab | Up to approximately 2 years

IPD SHARING:
Plan to Share IPD: No